CLINICAL TRIAL: NCT02378480
Title: A Phase 3 Randomized, Double-blind, Multi-center Study to Compare the Safety and Efficacy of Omadacycline IV/PO to Linezolid IV/PO for Treating Adults With Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: Omadacycline Versus Linezolid for the Treatment of ABSSSI (EudraCT #2013-003644-23)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-ABSI-1108
Record Dates: First submitted 2015-02-19; First posted 2015-03-04 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Bacterial Infections; Skin Structures and Soft Tissue Infections
MeSH Terms: conditions — Bacterial Infections; Soft Tissue Infections | interventions — omadacycline; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omadacycline (Experimental): Omadacycline IV; Omadacycline tablets
  Interventions: Drug: Omadacycline
- Linezolid (Active Comparator): Linezolid IV; Linezolid tablets
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Omadacycline — Injection for IV dosing; Tablets for oral dosing
  Arms: Omadacycline
Drug: Linezolid — Infusion solution for IV dosing; Tablets for oral dosing
  Other Names: Zyvox
  Arms: Linezolid

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of omadacycline as compared to linezolid in the treatment of adults with acute bacterial skin and skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ages 18 years or older who have signed the informed consent
* Has a qualifying skin and skin structure infection
* Female patients must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Infections where the outcome is strongly influenced by factors other than protocol-defined treatment and procedures, that require antibacterial treatment for greater than 14 days
* Evidence of significant immunological disease
* Severe sepsis or septic shock
* Has a history of hypersensitivity or allergic reaction to any tetracycline or to linezolid
* Has received an investigational drug within past 30 days
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (18):
  - Site 261, Mobile, Alabama
  - Site 262, Chula Vista, California
  - Site 254, La Mesa, California
  - Site 258, Oceanside, California
  - Site 252, Santa Ana, California
  - Site 260, Santa Ana, California
  - Site 269, Stockton, California
  - Site 259, Miami, Florida
  - Site 264, West Palm Beach, Florida
  - Site 256, Augusta, Georgia
  - Site 253, Columbus, Georgia
  - Site 257, Springfield, Massachusetts
  - Site 268, Detroit, Michigan
  - Site 266, Butte, Montana
  - Site 263, Las Vegas, Nevada
  - Site 270, Somers Point, New Jersey
  - Site 273, Buffalo, New York
  - Site 255, Rapid City, South Dakota
- Bulgaria (5):
  - Site 104, Pleven
  - Site 102, Plovdiv
  - Site 105, Plovdiv
  - Site 103, Rousse
  - Site 101, Sofia
- Croatia (5):
  - Site 205, Slavonski Brod
  - Site 201, Zagreb
  - Site 203, Zagreb
  - Site 202, Zagreb
  - Site 204, Zagreb
- Greece (4):
  - Site 207, Athens
  - Site 211, Athens
  - Site 208, Thessaloniki
  - Site 209, Thessaloniki
- Hungary (4):
  - Site 110, Budapest
  - Site 111, Budapest
  - Site 114, Miskolc
  - Site 113, Szeged
- Israel (4):
  - Site 213, Holon
  - Site 219, Kfar Saba
  - Site 214, Nazareth
  - Site 216, Safed
- Latvia (5):
  - Site 122, Daugavpils
  - Site 123, Liepāja
  - Site 124, Rēzekne
  - Site 120, Riga
  - Site 121, Riga
- Peru (6):
  - Site 234, Cusco
  - Site 233, Lima
  - Site 236, Lima
  - Site 238, Lima
  - Site 239, Lima
  - Site 237, Trujillo
- Poland (5):
  - Site 130, Bydgoszcz
  - Site 133, Katowice
  - Site 131, Lodz
  - Site 134, Olsztyn
  - Site 132, Warsaw
- Romania (7):
  - Site 141, Bucharest
  - Site 142, Bucharest
  - Site 146, Bucharest
  - Site 144, Cluj-Napoca
  - Site 140, Craiova
  - Site 143, Târgu Mureş
  - Site 145, Timișoara
- South Africa (2):
  - Site 241, Benoni, Gauteng
  - Site 244, Thabazimbi, Limpopo
- Spain (2):
  - Site 222, Terrassa, Barcelona
  - Site 221, Barcelona, Catalonia
- Turkey (Türkiye) (2):
  - Site 247, Ankara
  - Site 246, Trabzon
- Ukraine (9):
  - Site 172, Dnipropetrovsk
  - Site 173, Dnipropetrovsk
  - Site 179, Kharkiv
  - Site 171, Kyiv
  - Site 170, Lviv
  - Site 174, Odesa
  - Site 175, Uzhhorod
  - Site 178, Vinnytsia
  - Site 176, Zaporizhia

REFERENCES:
- [Derived] Rodriguez GD, Warren N, Yashayev R, Chitra S, Amodio-Groton M, Wright K. Intravenous Versus Oral Omadacycline or Linezolid for Acute Bacterial Skin and Skin Infections: A post hoc Analysis of the OASIS Trials. Infect Dis Ther. 2024 Dec;13(12):2637-2648. doi: 10.1007/s40121-024-01057-3. Epub 2024 Oct 26. PMID 39461915
- [Derived] Vacalis S, Brunton S, Gindi J. Omadacycline in Skin Infections and Pneumonia: A Review of the Evidence. J Fam Pract. 2022 Jun;71(5 Suppl):S10-S21. doi: 10.12788/jfp.0424. PMID 35776862
- [Derived] Pai MP, Wilcox MH, Chitra S, McGovern PC. Safety and efficacy of omadacycline by BMI categories and diabetes history in two Phase III randomized studies of patients with acute bacterial skin and skin structure infections. J Antimicrob Chemother. 2021 Apr 13;76(5):1315-1322. doi: 10.1093/jac/dkaa558. PMID 33458763
- [Derived] Cornely OA, File TM Jr, Garrity-Ryan L, Chitra S, Noble R, McGovern PC. Safety and efficacy of omadacycline for treatment of community-acquired bacterial pneumonia and acute bacterial skin and skin structure infections in patients with mild-to-moderate renal impairment. Int J Antimicrob Agents. 2021 Feb;57(2):106263. doi: 10.1016/j.ijantimicag.2020.106263. Epub 2020 Dec 14. PMID 33326848
- [Derived] Abrahamian FM, Sakoulas G, Tzanis E, Manley A, Steenbergen J, Das AF, Eckburg PB, McGovern PC. Omadacycline for Acute Bacterial Skin and Skin Structure Infections. Clin Infect Dis. 2019 Aug 1;69(Suppl 1):S23-S32. doi: 10.1093/cid/ciz396. PMID 31367742
- [Derived] O'Riordan W, Green S, Overcash JS, Puljiz I, Metallidis S, Gardovskis J, Garrity-Ryan L, Das AF, Tzanis E, Eckburg PB, Manley A, Villano SA, Steenbergen JN, Loh E. Omadacycline for Acute Bacterial Skin and Skin-Structure Infections. N Engl J Med. 2019 Feb 7;380(6):528-538. doi: 10.1056/NEJMoa1800170. PMID 30726689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to enroll adult participants with Acute Bacterial Skin and Skin Structure Infection (ABSSSI) that was known or suspected to be due to a Gram-positive pathogen(s). Randomization was stratified across treatment groups by type of infection (wound infection, cellulitis/erysipelas, and major abscess) and geographic region.
Pre-assignment Details: Participants who met inclusion criteria and did not meet exclusion criteria were randomly assigned to a treatment group, and received their first dose of test article within 4 hours after randomization. All participants were expected to present with ABSSSI severe enough to require a minimum of at least 3 days of intravenous treatment.
Groups:
- Omadacycline: Participants received intravenous (IV) omadacycline 100 milligrams (mg) every 12 hours (q12h) (2 doses), followed by 100 mg IV every 24 hours (q24h) (starting 24 hours after the first dose), with the option to switch to a 300 mg oral administration q24h after a minimum of 3 days (6 doses) of IV treatment (6 overall IV doses because of the blinding). Participants received 4 active doses plus 2 placebo doses to maintain the blind. The total treatment duration was 7 to 14 days.
- Linezolid: Participants received linezolid 600 mg IV q12h with the option to switch to a 600 mg oral administration q12h after a minimum of 3 days (6 doses) of IV treatment. The total treatment duration was 7 to 14 days.
Period: Overall Study
Arm/Group | Omadacycline | Linezolid
Started | 329 | 326
Completed | 301 | 294
Not Completed | 28 | 32
Not completed — Physician Decision | 1 | 1
Not completed — Death | 1 | 2
Not completed — Randomized, but Not Treated | 6 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Missed EOT/PTE Visit | 1 | 2
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 10 | 18

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received test article
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Linezolid | Total
Number analyzed (Participants) | 323 | 322 | 645
Age, Customized [Count of Participants; unit: Participants]
  18-45 years | 146 | 154 | 300
  >45-65 years | 141 | 136 | 277
  >65 years | 36 | 32 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 109 | 229
  Male | 203 | 213 | 416
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 12
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 16 | 8 | 24
  White | 294 | 300 | 594
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Clinical Response
Description: Early clinical response is defined as clinical success, which is categorized as survival with at least a 20% reduction of acute bacterial skin and skin structure infection (ABSSSI) primary lesion size compared to Screening measurements, without receiving any rescue antibacterial therapy. An indeterminate classification is used for a response that could not be adequately inferred because the participant was not assessed because they withdrew consent, were lost to follow-up, or other specified reason.
Time Frame: Screening; 48 to 72 hours after the first dose of test article
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants without a baseline sole Gram-negative ABSSSI pathogen
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 316 | 311
Participants
  Clinical success | 268 | 266
  Clinical failure | 23 | 19
  Indeterminate | 25 | 26
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = -0.7, 95% CI 2-sided [-6.3 to 4.9] — The 95% confidence interval was constructed based on the Miettinen and Nurminen method without stratification. Treatment difference for a response of clinical success was calculated as omadacycline minus linezolid

2. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the mITT Population at the Post Therapy Evaluation (PTE) Visit
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; the infection was sufficiently resolved such that further antibacterial therapy was not needed. These participants may have had some residual changes related to infection requiring ancillary treatment. Clinical Failure was defined as meeting any of the following criteria: infection required additional treatment with alternative antibacterial therapy; participant received antibacterial therapy between the End-of-Treatment (EOT) Visit and the PTE Visit that may have been effective for the infection under study for a different infection from the one under study; unplanned major surgical intervention for the infection under study between the EOT and PTE Visits; participant died before evaluation. Indeterminate: clinical response to test article could not be adequately inferred.
Time Frame: Screening; 7 to 14 days after the last day of therapy
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 316 | 311
Participants
  Clinical success | 272 | 260
  Clinical failure | 20 | 27
  Indeterminate | 24 | 24
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 2.5, 95% CI 2-sided [-3.2 to 8.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With the Indicated Investigator Assessment of Clinical Response in the Clinically Evaluable-Post Therapy Evaluation (CE-PTE) Population
Description: At the PTE Visit the investigator indicated one of the following outcomes relating to the primary infection under study: Clinical Success: participant was alive; the infection was sufficiently resolved such that further antibacterial therapy was not needed. These participants may have had some residual changes related to infection requiring ancillary treatment. Clinical Failure was defined as meeting any of the following criteria: infection required additional treatment with alternative antibacterial therapy; participant received antibacterial therapy between the EOT Visit and the PTE Visit that may have been effective for the infection under study for a different infection from the one under study; unplanned major surgical intervention for the infection under study between the EOT and PTE Visits; participant died before evaluation.
Time Frame: Screening; 7 to 14 days after the last day of therapy
Population: CE-PTE Population: all participants in the mITT Population meeting additional pre-defined criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 269 | 260
Participants
  Clinical success | 259 | 243
  Clinical failure | 10 | 17
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Non-Inferiority — A non-inferiority margin of 10% was used for the analysis; treatment difference = 2.8, 95% CI 2-sided [-1.0 to 6.9] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With the Indicated Type of Adverse Event (AE)
Description: An AE is defined as any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given a test article or in a clinical study. The event does not need to be causally related to the test article or clinical study. A serious adverse event (SAE) is defined as an event that resulted in death, was life-threatening, required hospitalization or prolongation of an existing hospitalization, resulted in a persistent or significant disability or incapacity, resulted in cancer, or resulted in a congenital anomaly or birth defect. A treatment-emergent AE (TEAE) is defined as any AE that newly appeared, increased in frequency, or worsened in severity on or after the initiation of active test article. Vital sign measurements, electrocardiogram findings, and laboratory values classified as adverse events were included in the analysis. Data are presented as the number of participants with at least 1 of the event.
Time Frame: 0 to 37 days
Population: Safety Population: all randomized participants who received test article
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 323 | 322
Participants
  AE | 158 | 157
  TEAE | 156 | 147
  Drug-releated AE | 58 | 59
  Severe TEAE | 6 | 10
  Serious TEAE | 12 | 8
  Drug-related serious TEAE | 0 | 0
  Serious TEAE leading to death | 1 | 2
  TEAE leading to premature drug discontinuation | 6 | 7
  TEAE leading to premature discontinuation of study | 6 | 7
  TEAE leading to dose interruption | 2 | 0
  Serious TEAEs leading to drug discontinuation | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the signing of Informed Consent Form to the time of the Final Follow-up assessment (up to 30 to 37 days after the start of the first infusion of test article).
Description: Adverse events are reported for members of the Safety Population, comprised of all randomized participants who received test article. Safety assessments included clinical review of reported adverse events and serious adverse events (SAEs). Treatment-emergent adverse events, defined as events occurring after the first dose of active test article, are reported.
Arm/Group | Omadacycline | Linezolid
All-Cause Mortality (participants affected / at risk) | 1/323 | 2/322
Serious Adverse Events (participants affected / at risk) | 12/323 | 8/322
Other Adverse Events (participants affected / at risk) | 104/323 | 101/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=323) | Linezolid (N=322)
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Subcutaneous Abscess (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Drug Abuse (Psychiatric disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=323) | Linezolid (N=322)
Nausea (Gastrointestinal disorders) | 40 | 32
Vomiting (Gastrointestinal disorders) | 17 | 16
Diarrhea (Gastrointestinal disorders) | 7 | 10
Infusion site extravasation (General disorders) | 28 | 19
Subcutaneous abscess (Infections and infestations) | 16 | 19
Cellulitis (Infections and infestations) | 13 | 14
Wound infection (Infections and infestations) | 8 | 5
Alanine aminotransferase increased (Investigations) | 9 | 14
Aspartate aminotransferase increased (Investigations) | 8 | 12
Headache (Nervous system disorders) | 10 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.